CLINICAL TRIAL: NCT00853905
Title: The Effect of Intracameral Triesence (Triamcinolone Acetonide Injectable Suspension) on Ocular Inflammation After Trabeculectomy, Tube Shunt Implantation or Combined Trabeculectomy With Cataract Surgery
Brief Title: Will the Use of Triesence During Glaucoma Surgery Provide Lower Eye Pressure and Improve the Results of the Surgery?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Marlene Moster, MD, Attending Surgeon Wills Eye Institute; Professor Jefferson Medical College, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-827
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Glaucoma
Keywords: open angle glaucoma (POAG); angle closure glaucoma (PACG); pigmentary glaucoma; pseudoexfoliation glaucoma; neovascular glaucoma; traumatic glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Exfoliation Syndrome; Glaucoma, Neovascular | interventions — Triamcinolone; Hanks Balanced Salt Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1(Triesence) (Experimental): glaucoma surgery with 0.2cc Triesence adjunct.
  Interventions: Drug: Triesence
- Treatment 2 (balanced salt solution BSS) (Active Comparator): glaucoma surgery with balanced salt solution, the standard technique.
  Interventions: Drug: balanced salt solution BSS

INTERVENTIONS:
Drug: Triesence — At end of standard glaucoma surgery and the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure, 0.2cc of Triesence will be delivered into the anterior chamber through the previously created paracentesis wound.
  Other Names: triamcinolone acetonide injectable
  Arms: Treatment 1(Triesence)
Drug: balanced salt solution BSS — At end of standard glaucoma surgery, the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure.
  Other Names: balanced salt solution
  Arms: Treatment 2 (balanced salt solution BSS)

SUMMARY:
The investigators hypothesize that intracameral Triesence during glaucoma surgery will provide lower intraocular pressure through better control of ocular inflammation, thus leading to a more successful filtering procedure.

DETAILED DESCRIPTION:
Determine the efficacy and safety of intracameral Triesence in patients who undergo trabeculectomy, tube shunt, or combined cataract extraction, intra-ocular lens implantation and trabeculectomy with or without adjunctive mitomycin-C.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients requiring surgery (Trabeculectomy or Express Shunt; Trabeculectomy plus Phacoemulsification and Interocular Lens Implant; Baerveldt Tube; Ahmed Tube; Molteno Tube)
* primary open angle glaucoma
* primary angle-closure glaucoma
* pseudoexfoliation glaucoma
* pigmentary glaucoma
* traumatic glaucoma
* neovascular glaucoma

Exclusion Criteria:

* patients that are pregnant, nursing, or not using adequate contraception
* any other eye surgery except cataract surgery
* an infection, inflammation, or any abnormality preventing measurement of eye pressure
* enrolled in another investigational study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene R Moster, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koval MS, Moster MR, Freidl KB, Waisbourd M, Jain SG, Ichhpujani P, Myers JS, Pro MJ. Intracameral triamcinolone acetonide in glaucoma surgery: a prospective randomized controlled trial. Am J Ophthalmol. 2014 Aug;158(2):395-401.e2. doi: 10.1016/j.ajo.2014.04.027. Epub 2014 May 2. PMID 24794283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2009 to July 2011 at the Wills Eye Hospital
Groups:
- Treatment 1(Triesence): 0.2cc Triesence
  At end of standard glaucoma surgery and the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure, 0.2cc of Triesence will be delivered into the anterior chamber through the previously created paracentesis wound.
- Treatment 2 (Balanced Salt Solution BSS): glaucoma surgery with balanced salt solution, the standard technique.
  At end of standard glaucoma surgery, the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure.
Period: Overall Study
Arm/Group | Treatment 1(Triesence) | Treatment 2 (Balanced Salt Solution BSS)
Started | 37 | 40
Completed | 35 | 36
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — never had surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment 1(Triesence): 0.2cc Triesence
  Triesence: At the end of standard glaucoma surgery after the anterior chamber is reformed with balanced salt solution or viscoelastic to adequate intraocular pressure; 0.2cc of Triesence will be delivered into the anterior chamber through the previously created paracentesis wound
- Treatment 2 (Balanced Salt Solution BSS): glaucoma surgery with balanced salt solution, the standard technique used.
  balanced salt solution BSS: standard technique for glaucoma surgery . At the end of the case anterior chamber will be reformed with balanced salt solution to adequate intraocular pressure.
- Total: Total of all reporting groups
Arm/Group | Treatment 1(Triesence) | Treatment 2 (Balanced Salt Solution BSS) | Total
Number analyzed (Participants) | 37 | 40 | 77
Age, Continuous [Median (Full Range); unit: years] | 68 [47 to 88] | 69 [42 to 88] | 68.5 [42 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 17 | 23 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 23 | 39
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 37 | 40 | 77
Interocular Pressure (mmHg) [Median (Full Range); unit: mmHg] | 24.5 [13 to 40] | 23.8 [8.5 to 56] | 24.0 [8.5 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Intraocular pressure (IOP) was measured by applanation tonometry in millimeters of mercury (mmHg). Surgical success was determined if IOP was <21mmHg and 20% less than baseline IOP. Failure was defined as inability to meet criteria for success or IOP was less than 5mmHg.
Time Frame: 1 day, 1week, 1 month, 3 month and 6 month post-op visits
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Treatment 2 (Balanced Salt Solution BSS): balanced salt solution At end of standard glaucoma surgery, the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure.
Arm/Group | Treatment 1(Triesence) | Treatment 2 (Balanced Salt Solution BSS)
Number analyzed (Participants) | 37 | 40
mm Hg
  Day 1 | 16.1 [13.1 to 19.05] | 12.8 [10.7 to 15.0]
  Week 1 | 11.7 [9.1 to 14.5] | 11.8 [9.8 to 13.9]
  Month 1 | 16.1 [13.0 to 19.4] | 14.4 [12.2 to 16.8]
  Month 3 | 15.1 [12.2 to 18.4] | 12.8 [10.7 to 15.1]
  Month 6 | 14.6 [11.7 to 17.8] | 13.6 [11.5 to 16.0]

2. Secondary Outcome: Anterior Chamber Inflammation (Flare)
Description: Inflammation in the anterior chamber (called flare), is measured 10 times per eye using the flare meter, a non-invasive measurement. Flare meter measures inflammation in photon counts per millisecond (p/msec).
Time Frame: 1 month, 3 month and 6 month post-op visits
Measure: Mean (95% Confidence Interval); unit: photon counts per millisecond (p/msec)
Groups:
- Treatment 1(Triesence): 0.2cc Triesence At end of standard glaucoma surgery, the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure.
Arm/Group | Treatment 1(Triesence) | Treatment 2 (Balanced Salt Solution BSS)
Number analyzed (Participants) | 37 | 40
photon counts per millisecond (p/msec)
  Month 1 | 0.4 [-0.2 to 0.8] | 1.0 [0.6 to 1.4]
  Month 3 | 0.6 [0 to 1.1] | 0.4 [-0.1 to 0.9]
  Month 6 | 0.3 [-0.2 to 0.8] | 0.2 [-0.2 to 0.7]

3. Secondary Outcome: Bleb Appearance
Description: A bleb is a blister on the white part of the eye (sclera) intentionally formed during some glaucoma surgeries. The Indiana Bleb Appearance Grading Scale (IBAGS) measures the bleb appearance in elevation (height), extent and vascularity. The height range is flat, low, moderate and high with 0 to 3 units on a scale. Zero is a flat bleb and 3 is a high bleb. Elevated functioning blebs increase the success of glaucoma surgery.
Time Frame: 1 day, 1 week, 1 month, 3 month and 6 month post-op visits
Population: Bleb assessment by IBAGS was not obtained at all visits. Overall, 20 of 37 (Triesence) and 20 of 40 (BSS) blebs were measured.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Triesence (Treatment 1): 0.2cc Triesence At end of standard glaucoma surgery and the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure, 0.2cc of Triesence will be delivered into the anterior chamber through the previously created paracentesis wound.
- Balanced Salt Solution (BSS Treatment 2): balanced salt solution (BSS) At end of standard glaucoma surgery, the anterior chamber is reformed with balanced salt solution or viscoelastic to an adequate intraocular pressure.
Arm/Group | Triesence (Treatment 1) | Balanced Salt Solution (BSS Treatment 2)
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 | 1.7 [1.4 to 2.1] | 2.1 [1.7 to 2.5]
  Week 1 | 1.7 [1.4 to 2.1] | 1.9 [1.5 to 2.3]
  Month 1 | 2.2 [1.8 to 2.6] | 1.9 [1.5 to 2.3]
  Month 3 | 2.0 [1.6 to 2.4] | 1.8 [1.4 to 2.2]
  Month 6 | 1.9 [1.5 to 2.3] | 2.1 [1.6 to 2.5]

4. Secondary Outcome: Patient Comfort
Description: Questionnaire administered to capture feeling of dry eye. Dry eye was graded on a scale of absent, mild, moderate and severe with 0 to 3 units on a scale.
Time Frame: 1 day, 1 week, 1 month, 3 month and 6 month post-op visits
Measure: Mean (95% Confidence Interval); unit: Patient comfort questionnaire score
Arm/Group | Treatment 1(Triesence) | Treatment 2 (Balanced Salt Solution BSS)
Number analyzed (Participants) | 37 | 40
Patient comfort questionnaire score
  Day 1 | 0.3 [0.1 to 0.6] | 0.1 [-0.1 to 0.4]
  Week 1 | 0.6 [0.4 to 0.9] | 0.3 [0 to 0.5]
  Month 1 | 0.3 [0 to 0.5] | 0.6 [0.4 to 0.9]
  Month 3 | 0.4 [0.1 to 0.6] | 0.4 [0.2 to 0.7]
  Month 6 | 0.7 [0.4 to 0.9] | 0.7 [0.5 to 0.9]

5. Secondary Outcome: Ocular Hypotensive Medications
Description: Number of ocular hypotensive ophthalmic solutions (eye drops) needed, if any, to maintain lower eye pressure.
Time Frame: 1 week, 1 month, 3 month, and or 6 month post-op visits
Measure: Mean (95% Confidence Interval); unit: eye drops
Arm/Group | Treatment 1(Triesence) | Treatment 2 (Balanced Salt Solution BSS)
Number analyzed (Participants) | 37 | 40
eye drops
  Week 1 | 0.03 [0.0 to 0.16] | 0.06 [0.02 to 0.2]
  Month 1 | 0.1 [0.04 to 0.26] | 0.03 [0 to 0.17]
  Month 3 | 0.08 [0.02 to 0.23] | 0.22 [0.11 to 0.41]
  Month 6 | 0.22 [0.11 to 0.39] | 0.22 [0.11 to 0.41]

ADVERSE EVENTS:
Time Frame: surgery, day 1, 1 week, 1 month, 3 month, 6 month
Arm/Group | Treatment 1(Triesence) | Treatment 2 (Balanced Salt Solution BSS)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/40
Other Adverse Events (participants affected / at risk) | 8/37 | 10/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1(Triesence) (N=37) | Treatment 2 (Balanced Salt Solution BSS) (N=40)
IOP failure (Eye disorders) | 7 (7) | 8 (8) — IOP failed to drop 20% or less than a 5mmhg drop from original IOP; eye drops added
choroidals drained; A/C reformed (Eye disorders) | 1 (1) | 2 (2) — patient needed another glaucoma procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No